CLINICAL TRIAL: NCT02277483
Title: Efficacy and Safety of LAIS® Mites Sublingual Tablets in Patients Aged Over 60 Years Suffering From House Dust Mite-induced Allergic Rhino-conjunctivitis With/Without Asthma
Brief Title: Efficacy and Safety of LAIS® Mites Sublingual Tablets
Acronym: korLAIS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Hae-Sim Park, professor, Department alleric internal medicine, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MED-CT4-14-159
Record Dates: First submitted 2014-10-20; First posted 2014-10-29 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Allergic Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- active treatment (Active Comparator): LAIS® Mites Sublingual tablets + rescue medication
  Interventions: Drug: LAIS®
- control (No Intervention): Rescue medication

INTERVENTIONS:
Drug: LAIS® — 10 X 1,000 / twice a week
  Other Names: active treatment
  Arms: active treatment

SUMMARY:
Evaluation of the efficacy and safety of SLIT with LAIS® Mites Sublingual tablets compared to standard drug treatment in patients aged over 60 years suffering from house dust mite (HDM) induced allergic rhino-conjunctivitis with/without asthma.

DETAILED DESCRIPTION:
The Total combined score (TCS), taking into account the rhinoconjunctivitis total symptom score (RTSS) and the total rescue medication score (RTMS), in the maximum expected mites exposition period (V4-V5) For the RTSS and the RTMS, the daily values as determined by the patients in their diary card are collected during the observation period over 30 days. Then, the mean daily scores during that period are calculated for both parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients aged 60 years or more with a history of at least two years of house dust mite (HDM) induced allergic rhinitis and/or allergic rhinoconjunctivitis with or without mild to moderate controlled asthma upon exposure to house dust mite [From the Global Strategy for Asthma Management and Prevention, Global Initiative for Asthma (GINA) 2007.
2. Clinically relevant sensitization to mites.
3. Positive clinical history of allergy due to house dust mite (HDM), proven by- The majority of perennial clinical symptoms appearing mostly related to indoor mites allergens

   * Specific Immunoglobulin E reactivity to mites allergens (ImmunoCAP>0.35 Ku/L)
   * Positive skin prick test (wheal diameter> 3mm, negative control < 2mm)
4. Retrospective Total Symptom Score (RRTSS) referred to the previous winter season greater than or equal to 8
5. Compliance and ability of the patient to complete a diary card for self-evaluation of the symptoms and anti-symptomatic medication
6. Signed and dated patient's Informed Consent

Exclusion Criteria:

1. Simultaneous participation in other clinical trials
2. Previous immunotherapy with mite allergens or cross reacting allergens within the last 5 years
3. Ongoing immunotherapy with any allergen
4. Patients being in any relationship or dependency with the sponsor and/or investigator
5. Other reasons contra-indicating an inclusion into the trial according to the investigator's estimation (e.g. poor compliance, inability of the patient to understand study documents and instructions)
6. Predominant seasonal allergic rhinitis
7. Patients with clinically relevant sensitization to seasonal aero-allergens occurring during the study period may not be included. Also patients with clinically relevant sensitization to perennial allergens like animal dander may not be included
8. Uncontrolled asthma
9. Chronic asthma or emphysema, particularly with a forced expiratory volume <70% of the predicted value and /or <70% of the individual optimum value
10. Infections of the oral cavity with severe symptoms
11. Patients with Galactose-intolerance, Lactase-deficiency, Glucose-Galactose-malabsorption
12. Active tuberculosis
13. Generally inflammatory as well as severe acute and chronic inflammatory diseases
14. Irreversible secondary disorders at the target organ (e.g. emphysema, bronchiectasis)
15. Immune deficiency (for example induced by immunosuppressive drugs)
16. Physician diagnosed diseases of the liver, spleen, nervous system, thyroidal gland as well rheumatic diseases, based on an autoimmune mechanism,
17. Malignancy
18. Alcohol abuse as well as drug and / or medication abuse
19. Patients treated with contra-indicated drugs
20. Contra-indication for adrenalin (for example, acute or chronic symptomatic coronary heart disease, severe hypertension, hyperthyroidism)
21. Completed or ongoing long-term treatment with tranquilizer or psycho active drugs
22. Completed or ongoing treatment with anti-Specific Immunoglobulin E-antibody
23. Uncontrolled asthma according to GINA guideline criteria

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Total combined score (TCS) | up to 48 weeks
  TCS = rhinoconjunctivitis total symptom score (RTSS) and the total rescue medication score (RTMS)

SECONDARY OUTCOMES:
sublingual immunotherapy | up to 48weeks
  usage of the Total Rescue Medication Score (RTMS)

CONTACTS AND LOCATIONS:
Overall Officials: hae-sim park, professor, Principal Investigator — Department of internal medicine
Locations (1):
- Jung-Won Park, Seoul, South Korea